CLINICAL TRIAL: NCT04953026
Title: SLAP Injury of the Shoulder Joint: Application Value of Deep Learning in Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020458
Record Dates: First submitted 2021-06-29; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Superior Labrum From Anterior to Posterior Injuries
Keywords: artificial intelligence; SLAP; diagnosis
MeSH Terms: conditions — Shoulder Injuries; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal control group-Grade 0: Arthroscopic examination of the labrum was normal, and the labrum was intact without injury or tear.
  Interventions: Diagnostic Test: Diagnositic test
- Ligament injury -Grade 1: Arthroscopic examination of the shoulder showed labrum degeneration or injury, but no local or complete tear.
  Interventions: Diagnostic Test: Diagnositic test
- Ligament tear-Grade 2: Arthroscopy of the shoulder revealed partial or complete loss of labrum.
  Interventions: Diagnostic Test: Diagnositic test

INTERVENTIONS:
Diagnostic Test: Diagnositic test — The results of shoulder arthroscopy were taken as the gold standard, and MRI examination was taken as the research object.

SUMMARY:
This study intends to study the shoulder SLAP injury through deep learning technology and establish a deep learning model through the combination of axial and oblique coronal images to establish a deep learning method that can accurately identify and grade shoulder SLAP injury.

DETAILED DESCRIPTION:
1. Recognition of labrum images based on LeNet: axial and oblique coronal T2-fs images were used, and all images were corrected and standardized. LeNet identified the images with labrum of the shoulder joint, and the images with labrum structure of shoulder joint were selected from the complete sequence. In contrast, the images without labrum structure were deleted. All the data are divided into a training set (70%, 30% in training set as verification set), and the remaining 30% as a test set to evaluate the accuracy of model recognition. Enter the obtained results into the next step.
2. Recognition and segmentation of glenoid lip of shoulder joint based on DenseNet: the labrum is recognized by DenseNet in the selected image. The labelimg software based on Python was used to locate the labrum coordinates and then input them into Python for recognition learning. All the data were divided into a training set (70% and 30% of the training set were selected as the verification set). The remaining 30% was used as the test set to evaluate the accuracy of model recognition. After identifying the labrum structure, the labrum structure is locally cut and enlarged to remove the redundant information and improve the recognition efficiency and accuracy. Finally, input the result to the next step.
3. Recognition and grading of shoulder SLAP injury based on 3D-CNN: recognition and grading of input data through 3D-CNN model. 3D-CNN is divided into eight layers: input layer, hard wire layer H1, convolution layer C2, downsampling layer S3, convolution layer C4, downsampling layer S5, convolution layer C6 and output layer. 3D-CNN constructs a cube by stacking multiple consecutive frames and then uses a 3D convolution kernel in the cube. Through this structure, the feature images in the convolution layer will be connected with multiple adjacent frames in the previous layer to realize the information acquisition of continuous images. Similarly, the data is divided into a training set (70%, and then 30% of the training set is selected as the verification set), and the remaining 30% is used as the test set to evaluate the classification accuracy to identify whether there is labrum injury and grade the image with injury.
4. Establish CNN combined model: after establishing the model for the axial and oblique coronal view according to the above process (1-3), according to the output characteristics of the CNN classification model, predict the probability of different grades before the output results, and the output results are based on these probabilities to select the expression form of the maximum possible probability. Our combined model averages the probabilities of these different classifications, calculates the final prediction probability, and then obtains the final joint model. The test set of the third step (including the mixed data of axial and coronal images) was used to verify the joint model.

ELIGIBILITY:
Inclusion Criteria:

1. Without any treatment before imaging examination;
2. MR of the shoulder joint was performed within 3 months before the operation and the image quality was good;
3. Arthroscopic operation was performed in our hospital, and the operation records were complete.

Exclusion Criteria:

1. History of shoulder surgery, tumor, or previous fracture;
2. Unclear image, serious artifact, or incomplete clinical data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Collect and analyze patients who underwent shoulder MR examinations in the Department of Radiology, Peking University Third Hospital from September 2018 to September 2020.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
SLAP Injury of the Shoulder Joint: Application Value of Deep Learning in Diagnosis | 2021.10.1-2022.7.1
  The model of deep learning was obtained for diagnosis and grading of SLAP injury and compared with the radiologists of different stages.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No